CLINICAL TRIAL: NCT07347340
Title: Effectiveness Of Bushen Tongzhi Formula Pretreatment On Pregnancy Outcomes In Infertile Women With Diminished Ovarian Reserve Undergoing In Vitro Fertilization And Embryo Transfer: Study Protocol For A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial (PRIME Study)
Brief Title: Testing Herbal Pretreatment For IVF Success In Women With Low Ovarian Reserve
Acronym: PRIME
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K9218; 2025-PUMCH-C-020 (Other Grant/Funding Number: National High Level Hospital Clinical Research Funding)
Record Dates: First submitted 2025-12-24; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Diminished Ovarian Reserve (DOR)
Keywords: Traditional Chinese Medicine; Bushen Tongzhi Formula; Diminished Ovarian Reserve; Infertility; In Vitro Fertilization; Randomized Controlled Trial; Multicenter Study; Herbal Medicine; Adjuvant Therapy; Ovarian Response; Pregnancy Rate; Kidney Deficiency; Chinese Medicine Pattern; PRIME Study
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Parallel Assignment. Participants are randomly assigned to one of two treatment groups (herbal formula or placebo) in a 1:1 ratio and remain in that group for the duration of the intervention.
  Triple (Participant, Care Provider, Outcomes Assessor). The study is double-blind, meaning neither the participants nor the investigators know the treatment assignment. Outcomes assessors (e.g., embryologists, sonographers) are also blinded. This is achieved using a matched, indistinguishable placebo.
  The primary purpose is Treatment, to evaluate the efficacy of the herbal intervention compared to placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The data manager and the statistician performing the interim and primary analyses are also masked to group assignment until after the database is locked for the final analysis. This ensures blinding is maintained throughout the data processing and analysis phases to prevent bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bushen Tongzhi Formula Pretreatment plus Standard IVF/ICSI (Experimental): Intervention: Participants in this arm receive the investigational treatment, which consists of oral administration of the Bushen Tongzhi Formula granules combined with a standard IVF/ICSI protocol.
  Details:
  Medication: "Bushen Tongzhi Formula" herbal granules (20g per dose).
  Dosage & Administration: 20g (one sachet), taken orally three times daily after meals.
  Treatment Regimen: The intervention includes a 3-month pretreatment phase prior to the start of ovarian stimulation. Participants continue taking the medication concurrently throughout their subsequent IVF/ICSI treatment cycle (including during gonadotropin stimulation and until pregnancy confirmation). The maximum total treatment duration is 6 months, stopping upon confirmation of clinical pregnancy.
  Concurrent Procedure: All participants undergo a standard, clinic-determined controlled ovarian stimulation protocol for IVF or ICSI, followed by egg retrieval, embryo culture, and fresh or frozen-thawed embryo transfer.
  Interventions: Drug: Bushen Tongzhi Formula
- Placebo Pretreatment plus Standard IVF/ICSI (Placebo Comparator): Intervention: Participants in this arm receive the control treatment, consisting of an oral placebo combined with a standard IVF/ICSI protocol.
  Details:
  Medication: Matched placebo granules. These contain no active herbal ingredients and are formulated from inert materials (e.g., dextrin, food-grade flavorings/colorants) to precisely mimic the appearance, taste, smell, and packaging of the active Bushen Tongzhi Formula granules.
  Dosage & Administration: 20g (one sachet), taken orally three times daily after meals.
  Treatment Regimen: The regimen is identical to the experimental arm: a 3-month pretreatment phase, followed by continued placebo intake concurrently throughout the subsequent IVF/ICSI treatment cycle. The maximum total duration is 6 months, with medication stopping upon confirmation of clinical pregnancy.
  Concurrent Procedure: Participants undergo the same standard, clinic-directed IVF/ICSI procedures.
  Interventions: Drug: Placebo Pretreatment plus Standard IVF/ICSI

INTERVENTIONS:
Drug: Bushen Tongzhi Formula — Bushen Tongzhi Formula is a standardized, fixed-composition herbal formula developed based on Traditional Chinese Medicine (TCM) principles for treating diminished ovarian reserve due to kidney deficiency. It is composed of multiple herbal ingredients processed into a granulated formulation. The dosage is 20g of granules taken orally three times daily. It serves as the active comparator against an indistinguishable placebo in this trial.
  Arms: Bushen Tongzhi Formula Pretreatment plus Standard IVF/ICSI
Drug: Placebo Pretreatment plus Standard IVF/ICSI — Intervention: Participants in this arm receive the control treatment, consisting of an oral placebo combined with a standard IVF/ICSI protocol.
  Details:
  Medication: Matched placebo granules. These contain no active herbal ingredients and are formulated from inert materials (e.g., dextrin, food-grade flavorings/colorants) to precisely mimic the appearance, taste, smell, and packaging of the active Bushen Tongzhi Formula granules.
  Dosage & Administration: 20g (one sachet), taken orally three times daily after meals.
  Treatment Regimen: The regimen is identical to the experimental arm: a 3-month pretreatment phase, followed by continued placebo intake concurrently throughout the subsequent IVF/ICSI treatment cycle. The maximum total duration is 6 months, with medication stopping upon confirmation of clinical pregnancy.
  Concurrent Procedure: Participants undergo the same standard, clinic-directed IVF/ICSI procedures.
  Arms: Placebo Pretreatment plus Standard IVF/ICSI

SUMMARY:
The goal of this clinical trial is to learn if a traditional Chinese herbal pretreatment can improve pregnancy outcomes in infertile women with diminished ovarian reserve (DOR) who are undergoing in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI). The main question it aims to answer is:

• Does pretreatment with the Bushen Tongzhi Formula increase the cumulative clinical pregnancy rate from a single egg retrieval cycle compared to a placebo?

Researchers will compare the group taking the herbal formula to the group taking a placebo to see if the herbal formula is more effective.

Participants will:

* Take the assigned study medication (herbal formula or placebo) three times daily for 3 months before starting IVF/ICSI.
* Continue taking the medication during their IVF/ICSI treatment cycle, for up to 6 months total.
* Undergo standard IVF/ICSI procedures as planned by their doctor.
* Have their pregnancy outcomes and health monitored through clinic visits and their medical records.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, superiority clinical trial. The study aims to evaluate the efficacy and safety of a standardized traditional Chinese medicine (TCM) formula, the "Bushen Tongzhi Formula" (also referred to as the "Xiehe DOR Bushen Tongzhi Formula"), as a pretreatment and adjuvant therapy in infertile women with Diminished Ovarian Reserve (DOR) undergoing in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI).

Background DOR, characterized by a reduced quantity and/or quality of oocytes, presents a significant challenge in assisted reproductive technology (ART), often leading to poor ovarian response, fewer retrievable oocytes, and lower pregnancy rates. While controlled ovarian stimulation protocols continue to evolve, there remains a critical need for interventions that can improve ovarian function and oocyte quality prior to ART cycles. TCM, guided by the theory of "the kidney governing reproduction," offers a potential approach by addressing the root pattern of "kidney essence deficiency," which is central to DOR in TCM diagnostics. Preliminary observations of the Bushen Tongzhi Formula have suggested potential benefits, but robust evidence from large-scale, rigorously designed trials is lacking.

Study Population The study will enroll 348 infertile female participants, aged 22 to 39 years, diagnosed with DOR according to standardized criteria (requiring at least two of the following: baseline FSH 10-25 IU/L, AMH <1.1 ng/mL, or antral follicle count <7). All participants must also meet TCM diagnostic criteria for Kidney Deficiency pattern and be planning to undergo a fresh IVF/ICSI cycle. Key exclusions include significant uterine abnormalities, known chromosomal disorders, severe medical or psychiatric conditions, active genital infections, advanced endometriosis, plans for donor egg or PGT cycles, and a history of multiple prior IVF failures.

Interventions Eligible participants will be randomly assigned in a 1:1 ratio via a centralized interactive web response system (IWRS), stratified by study site and age.

Experimental Group: Participants will take the Bushen Tongzhi Formula granules (20g, three times daily) for a 3-month pretreatment phase. Upon starting their standardized IVF/ICSI protocol, they will continue the herbal medication concurrently for up to an additional 3 months, stopping upon confirmation of clinical pregnancy. The maximum total treatment duration is 6 months.

Control Group: Participants will follow an identical regimen but will take a matched placebo granules that are indistinguishable from the active drug in appearance, taste, and packaging.

Both groups will receive standard lifestyle counseling and undergo the same clinic-directed IVF/ICSI protocols, including gonadotropin stimulation, trigger, egg retrieval, fertilization, and embryo transfer.

Outcomes The primary outcome is the cumulative clinical pregnancy rate resulting from a single egg retrieval cycle (including fresh and subsequent frozen embryo transfers from that cycle).

Secondary outcomes encompass multiple dimensions:

Ovarian Response: Gonadotropin dose/duration, number of oocytes retrieved, MII oocyte rate, cycle cancellation rate.

Embryological Outcomes: Fertilization rate, cleavage rate, high-quality embryo rate, blastocyst formation rate.

Endometrial Receptivity: Endometrial thickness and pattern on day of trigger/transfer.

Pregnancy & Neonatal Outcomes: Biochemical pregnancy, ongoing pregnancy, miscarriage, ectopic pregnancy, and live birth rates; neonatal birth weight and major malformations.

TCM Efficacy: Change in Kidney Deficiency symptom score.

Safety: Incidence and severity of adverse events (AEs) and serious AEs (SAEs); changes in vital signs, body mass index, and laboratory parameters (hematology, liver and kidney function).

Study Procedures & Data Collection The study employs a pragmatic, integrated data collection strategy to minimize participant burden. Key efficacy and safety data are captured at predefined visits (V0-V9) spanning screening, treatment, and pregnancy follow-up. Crucially, data from routine ART procedures (egg retrieval, embryology, pregnancy tests, ultrasound scans) are extracted by trained staff from hospital electronic medical records and laboratory systems, eliminating the need for extra visits solely for research purposes. Post-intervention pregnancy and neonatal outcomes are collected via medical record review and structured telephone interviews at 42 days and 6 months postpartum.

Statistical Analysis The sample size of 348 participants (174 per group) was calculated to detect an absolute 15% improvement in the cumulative clinical pregnancy rate (from 25% in the control group to 40% in the experimental group) with 80% power and a one-sided alpha of 0.025, accounting for a 15% dropout rate. The primary analysis will be performed on the Full Analysis Set (intent-to-treat principle) using the Cochran-Mantel-Haenszel test, controlling for study site. A superiority conclusion will be reached if the lower bound of the 95% confidence interval for the difference in rates is greater than zero and the p-value is <0.025. Secondary continuous and categorical outcomes will be analyzed using ANCOVA (adjusted for baseline) and appropriate chi-square tests, respectively. Safety will be analyzed in the Safety Set.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 22 to 39 years (inclusive).
* Diagnosis of diminished ovarian reserve (DOR), defined by meeting at least two of the following three criteria: 1, Basal follicle-stimulating hormone (FSH) level between 10 and 25 IU/L (measured on menstrual cycle days 2-4); 2, Anti-Müllerian hormone (AMH) level < 1.1 ng/mL; 3, Antral follicle count (AFC) < 7 (total count of follicles 2-10 mm in diameter in both ovaries).
* Diagnosis of infertility, defined as failure to achieve a clinical pregnancy after 12 months or more of regular unprotected sexual intercourse.
* Diagnosis of Kidney Deficiency pattern according to Traditional Chinese Medicine criteria, as defined in the study protocol.
* Scheduled to undergo a fresh in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) cycle.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Uterine structural abnormalities likely to impair implantation or pregnancy (e.g., untreated submucosal fibroids, severe intrauterine adhesions, uterine septum).
* Known abnormal karyotype in either partner.
* Uncontrolled or severe medical conditions (e.g., hypertension, diabetes, thyroid dysfunction, hepatic/renal insufficiency, symptomatic heart disease).
* Diagnosed severe psychiatric disorders (e.g., schizophrenia, bipolar disorder).
* History of prior pelvic radiation or cytotoxic chemotherapy.
* Active genital tract infection.
* Diagnosed or suspected severe (ASRM stage III-IV) endometriosis with recurrent symptoms.
* Planned use of donor oocytes or preimplantation genetic testing (PGT).
* History of repeated IVF/ICSI failure (≥3 failed egg retrieval cycles or ≥3 failed transfers of high-quality embryos).
* Known allergy to any component of the investigational herbal formula.
* Participation in another clinical trial within the past 3 months.
* Use of medications known to affect ovarian function (e.g., DHEA, growth hormone) within the past month.
* Current heavy alcohol consumption or smoking.
* Any other condition deemed by the investigator to make the participant unsuitable for the study.

Ages: 22 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 348 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative clinical pregnancy rate from a single oocyte retrieval cycle | From randomization until 12 months after the oocyte retrieval procedure.
  This outcome measures the proportion of participants in each treatment group who achieve a clinical pregnancy resulting from a single oocyte retrieval procedure. A clinical pregnancy is defined as the ultrasound confirmation of an intrauterine gestational sac with cardiac activity. The rate is "cumulative" because it includes pregnancies achieved from both the initial fresh embryo transfer and any subsequent frozen-thawed embryo transfer(s) utilizing all embryos derived from that single retrieval cycle. Data will be collected until no embryos from the index cycle remain for transfer or a clinical pregnancy is confirmed.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) from this trial is not currently planned for public sharing due to strict patient privacy regulations under Chinese law and institutional data governance policies. The data contains sensitive personal health information. Future sharing of de-identified data may be considered for specific collaborative research purposes upon formal request and approval by the study's steering committee, contingent on compliance with data transfer agreements and ethical review.